CLINICAL TRIAL: NCT03298763
Title: Targeted Stem Cells Expressing TRAIL as a Therapy for Lung Cancer
Acronym: TACTICAL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: UCL/14/0453
Record Dates: First submitted 2017-09-20; First posted 2017-10-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Adenocarcinoma of Lung
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Intervention Model Description: Phase I:
  Single centre, accelerated dose dose de-escalation design with a modified Bayesian continual reassessment method (mCRM) to estimate the recommended Phase II dose (RP2D) of MSCTRAIL in combination with pemetrexed/cisplatin chemotherapy.
  Phase II:
  Multicentre, randomised double blind placebo controlled trial comparing MSCTRAIL at the RP2D and pemetrexed/cisplatin chemotherapy versus pemetrexed/cisplatin chemotherapy alone.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 - RP2D finding study (Experimental): Phase I of the trial aims to establish the recommended MSCTRAIL dose when given in combination with cisplatin/pemetrexed chemotherapy in metastatic non-small cell lung cancer (NSCLC) patients
  Interventions: Genetic: MSCTRAIL
- Phase 2 Intervention Arm (Active Comparator): Cisplatin 75mg/m2 and Pemetrexed 500mg/m2 on day 1 followed by MSCTRAIL (at the recommended phase 2 dose) on day 2. This schedule will be repeated after 21 days for 3 cycles.
  Patients will then receive a further 1-3 cycles of pemetrexed/ cisplatin alone. They may then be eligible for maintenance pemetrexed according to clinical response as directed by their Oncologist in line with local standard of care.
  Interventions: Genetic: MSCTRAIL
- Phase 2 Control Arm (Placebo Comparator): cisplatin 75mg/m2 and pemetrexed 500mg/m2 on day 1 and placebo on day 2. This will be repeated after 21 days for up to 3 cycles.
  Patients will then receive a further 1-3 cycles of pemetrexed/ cisplatin alone. They may then be eligible for maintenance pemetrexed according to clinical response as directed by their Oncologist in line with local standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Genetic: MSCTRAIL — 3 doses of MSCTRAIL, administered as an intravenous 60 minutes infusion over 3 cycles, in combination with standard chemotherapy (Cisplatin/Pemetrexed).
  After 3 cycles patients will have 1-3 further treatment of pemetrexed and cisplatin without MSCTRAIL.
  Other Names: Mesenchymal stromal cells genetically modified to express TRAIL
  Arms: Phase 1 - RP2D finding study; Phase 2 Intervention Arm
Drug: Placebo — Placebo will be made up of the same material used to cryopreserve the ATIMP (MSCTRAIL) but will not include the active product
  Arms: Phase 2 Control Arm

SUMMARY:
The aim of the study is to evaluate the safety and anti-tumour activity of MSCTRAIL in addition to chemotherapy in metastatic Non-small cell lung cancer (NSCLC) patients in a Phase I/II clinical trial.

In the phase I study, patients will receive cisplatin and pemetrexed on day one followed by MSCTRAIL cells on day 2. This constitutes one cycle of treatment. Each patient will receive 3 cycles of treatment at 21 day intervals. The aim of phase 1 is to estimate the recommended Phase II dose (RP2D) of MSCTRAIL in combination with pemetrexed/cisplatin chemotherapy.

During the phase II study patients will be randomised to either the intervention or the control arm of the study. All patients in both arms will receive cisplatin and pemetrexed on day one of treatment. Patients randomised to the intervention arm will receive the recommended dose of MSCTRAIL from Phase I on day 2 whilst those in the control arm will receive a placebo. As this is a double blind trial both patients and the clinical team will not know whether they are receiving MSCTRAIL or a placebo product. The aim of phase 2 is to assess tolerability and preliminary efficacy of MSCTRAIL in combination with pemetrexed/cisplatin chemotherapy.

DETAILED DESCRIPTION:
Phase 1:

A first-in-human, single-centre, accelerated, dose de-escalation design with a modified Bayesian continual reassessment method (mCRM) to estimate the recommended Phase II dose (RP2D) of MSCTRAIL in combination with pemetrexed/cisplatin chemotherapy.

The first cohort of three patients will receive cisplatin 75mg/m2 and pemetrexed 500mg/m2 on day 1 followed by the highest dose of MSCTRAIL, 4x10^8 cells, on day 2. This schedule will be repeated every 21 days until 3 cycles of treatment have been delivered. It is expected that patients will receive 4-6 cycles of cisplatin/pemetrexed in total and may continue with maintenance pemetrexed thereafter.

If there are no DLTs within the first cohort then a subsequent expansion cohort will receive the same regimen of cisplatin/pemetrexed and MSCTRAIL and data from this expansion cohort will be used to determine the recommended phase 2 dose (RP2D). Between 6 and 12 patients will be enrolled into phase I of the trial depending on the number of cohorts assessed.

Phase 2:

A multicentre, randomised, placebo controlled trial comparing MSCTRAIL at the RP2D and pemetrexed/cisplatin chemotherapy versus pemetrexed/cisplatin chemotherapy alone.

Patients will be randomised 1:1 between the intervention and control arm. Patients entering the intervention arm will receive cisplatin 75mg/m2 and pemetrexed 500mg/m2 on day 1 followed by MSCTRAIL at the RP2D on day 2. This schedule will be repeated after 21 days for 3 cycles.

Patients in the control arm with receive cisplatin 75mg/m2 and pemetrexed 500mg/m2 on day 1 and placebo on day 2. This will be repeated after 21 days for up to 3 cycles.

At this point patients will receive a further 1-3 cycles of pemetrexed/ cisplatin alone. They may then be eligible for maintenance pemetrexed according to clinical response as directed by their Oncologist in line with local standard of care.

ELIGIBILITY:
1. Inoperable stage IIIb/IV histologically/cytologically confirmed lung adenocarcinoma
2. EGFR mutation and EML4-ALK translocation negative
3. Patients with evaluable but unmeasurable disease can be included in the phase I study, but disease must be measurable (CT scan must be within 28 days of randomisation) to be included in the phase II study
4. ECOG performance status of 0 or 1
5. Life expectancy of at least 12 weeks
6. Age at least 18 years
7. Adequate haematological status:

   1. Haemoglobin ≥100g/L
   2. Neutrophil count ≥1.5 x 109/L
   3. Platelets ≥100 x 109 /L
8. Adequate organ function:

   1. Bilirubin ≤1.5 x ULN
   2. ALT or AST ≤3 x ULN (≤5 x ULN is acceptable with liver metastases)
   3. Creatinine clearance ≥ 60 ml/min (C&G or EDTA)
9. Negative pregnancy test for female patients of child bearing potential.
10. Male subjects and women of child bearing potential must agree to use an acceptable method of birth control for the duration of the trial and for 12 months after the last trial treatment administration.
11. Ability to understand and provide written informed consent
12. Ability to comply with the requirements of the protocol

Exclusion Criteria:

1. Prior chemotherapy, hormonal therapy, radiotherapy (including palliative radiotherapy), immunotherapy or treatment with an investigational drug for advanced NSCLC.
2. Any surgical procedure in the previous 6 weeks prior to registration/ randomisation
3. Known respiratory failure with baseline resting SpO2 <88%
4. Long term oxygen therapy
5. Severe intercurrent infection
6. Active or infected wounds
7. Yellow fever vaccination within 30 days prior to trial registration/randomisation
8. Subject has known sensitivity to any of the trial drugs to be administered during the trial.
9. Any contraindication to the administration and use of cisplatin, pemetrexed, vitamin B12 or folic acid
10. Prior malignancy other than NSCLC (except if the tumour was a non-melanoma skin tumour that has been completely excised or in situ cervix carcinoma), unless have been treated with curative intent with no evidence of disease for > 3 years
11. Evidence of symptomatic brain metastases requiring treatment
12. Myocardial infarction, or unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure [New York Heart Association > class II]) within 1 year of enrolment
13. Known inflammatory bowel disease
14. Known hepatitis B or C infection, human immunodeficiency virus (HIV)-positive patients
15. Pregnant women or those who are breast feeding
16. Other medications, severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, or may interfere with the interpretation of trial results, and in the judgment of the investigator would make the patient inappropriate for entry into this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Determination of recommended Phase II dose (RP2D) of MSCTRAIL in combination of cisplatin and pemetrexed treatment (Phase 1) | until 21 days after the last dose of MSCTRAIL
  The dose recommended for phase II (i.e. the Maximum Tolerated Dose, or MTD) will be the largest dose that has an estimated risk of causing DLT (defined as MSCTRAIL related adverse event of grade 3 or higher) equal or closest to the target level of 35% (the target toxicity level). A modified Bayesian continual reassessment method (mCRM) will be used.
Tumour response rate (Phase 2) | 12 weeks post 1st MSCTRAIL infusion
  At each visit patients will be assigned a RECIST visit response of CR, PR, SD or PD depending on the status of their disease compared to baseline and previous assessments.
  Objective tumour response rate is defined as the percentage of patients who have a confirmed visit response of CR or PR prior to any evidence of progression (as defined by RECIST 1.1).

SECONDARY OUTCOMES:
Frequency of adverse events (Phase 1 & 2) | Up to 12 weeks post 1st MSCTRAIL infusion
  Adverse events (AEs) will be listed individually by patient and dose group (dose and schedule). The number of patients experiencing each AE will be summarised by the CTCAE grade. The number and percentage of patients with adverse events in different categories (eg, causally related, CTCAE grade ≥3 etc) will be summarised by dose group, and events in each category will be further summarised.
Best Overall response (Phase 1&2) | Until end of follow up period (Phase 1: 1 year post last treatment, Phase 2: 2 years post last treatment)
  Tumour response data will be summarised using the following response categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD) and Non-Evaluable (NE).
  Waterfall plots (bar charts) indicating the percentage change from baseline in sum of the diameters of target lesions (TLs) may be produced depending on how much data is obtained in patients with measurable disease at baseline. These may be individual patient plots of changes in tumour size over time or dose level plots with the best percentage change per patient displayed.
Progression free survival (Phase 1 & 2) | End of follow up period (Phase 1: 1 year post last treatment, Phase 2: 2 years post last treatment)
  Progression Free Survival (PFS) is defined as the time from randomization to time of progression (as per RECIST v1.1 criteria) or time of death from any cause. PFS will be analysed using KM plots and will be presented along with median PFS.
Overall survival (Phase 2) | End of follow up period (2 years post last treatment)
  Overall Survival (OS) is defined as the time from randomization to time of death from any cause. OS will be analysed using KM plots and will be presented along with median OS.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Janes, Principal Investigator — UCL
Locations (1):
- University College London Hospital, London, United Kingdom